CLINICAL TRIAL: NCT04149158
Title: Evaluation of Sinetrol® Xpur in Fat Mass Reduction on Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNTCT2015
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Change in Total Body Fat Mass Percentage Loss Versus Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Verum (Experimental): Sinetrol® Xpur
  Interventions: Dietary Supplement: Sinetrol® Xpur

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Sinetrol® Xpur
  Arms: Verum

SUMMARY:
This study aims to evaluate effects of a 16-week supplementation with a polyphenol rich extract, Sinetrol® Xpur, on fat mass accumulation and body weight management improvement.Subjects were overweight or obese and received polyphenol supplement or placebo. A 4-week follow-up as performed to evaluate its effect after supplementation stop.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (25 kg.m-2<BMI<42.5kg.m-2)
* healthy

Exclusion Criteria:

* metabolic or chronical disease with treatments (i.e.: diabetes, dyslipidemia, thyroiditis, inflammatory disease, immunological disease, infectious disease, asthma, anxiety and depression)
* food allergy to the ingredients of the product (grapefruit, orange, caffeine, guarana)
* involved in the prior 6 months in a chronic treatment program, eating disorders history, subjected to weight reduction by surgery
* start or quit smoking, high alcohol consumption
* pregnant, breastfeeding, wanting to have a baby,
* menopausal women

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — stratification of sex (40%minimum and 60% maximum of each sex)
Enrollment: 77 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in total body fat percentage loss versus bodyweight | week1; week16; week20

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alcaraz Ramon, Principal Investigator — UCAM
Locations (1):
- UCAM, Murcia, Spain

REFERENCES:
- [Derived] Muralidharan J, Romain C, Martinez-Noguera FJ, Marin-Cascales E, Chung L, Alcaraz P, Cases J. A 16-week supplementation with a polyphenol-rich supplement, Sinetrol(R) Xpur, aids in fat loss of overweight and obese volunteers: a randomised, double-blind, parallel trial. Int J Food Sci Nutr. 2026 Feb;77(1):40-47. doi: 10.1080/09637486.2025.2589845. Epub 2025 Dec 15. PMID 41399165